CLINICAL TRIAL: NCT05684848
Title: Interventional Pilot Study to Evaluate the Effect of a Resveratrol-based Nasal Spray Associated With Carboxymethylbetaglucan in Isotonic Solution in the Prevention of RTI in Children With Pre-school Wheezing
Brief Title: Evaluate the Effect of Nasal Spray in the Prevention of RTI in Children With Pre-school Wheezing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Noos S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LFV_PRE
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Wheezing; Recurrent Respiratory Tract Infections
Keywords: RRI; Wheezing; Medical Device; Resveratrol
MeSH Terms: conditions — Respiratory Sounds; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol + CMG (Active Comparator): Medical device: nasal spray based on resveratrol associated with carboxymethylbetaglucan in isotonic solution
  Interventions: Device: Resveratrol + CMG
- Isotonic solution (Placebo Comparator): Medical Device with isotonic solution
  Interventions: Device: Isotonic solution

INTERVENTIONS:
Device: Resveratrol + CMG — As prevention (resveratrol or its placebo) 2 puffs per nostril 2 times a day (morning and evening) for a period of 3 months. If during the preventive administration of the spray the first symptoms of a viral infection should appear, the parent should increase the dosage of the nasal spray to 2 puffs per nostril 4 times a day.
  Arms: Resveratrol + CMG
Device: Isotonic solution — As prevention (resveratrol or its placebo) 2 puffs per nostril 2 times a day (morning and evening) for a period of 3 months. If during the preventive administration of the spray the first symptoms of a viral infection should appear, the parent should increase the dosage of the nasal spray to 2 puffs per nostril 4 times a day.
  Arms: Isotonic solution

SUMMARY:
To determine whether or not preventive administration of resveratrol in the form of a nasal spray is effective in reducing the number of asthma exacerbations typical of preschool wheezing children who develop viral infections.

DETAILED DESCRIPTION:
The surface of the mucous membranes represents the first gateway for many viral agents including respiratory and intestinal ones which have the greatest epidemiological value. Viruses cause damage to these epithelia and can favor bacterial superinfection as well as complications of already existing pathologies; it is therefore essential to identify non-toxic substances that can hinder the entry of the virus and consequently its replication.

Both wheezing and viral infections are common in children, especially under the age of five. In fact, it is recorded that around 25% of children within nine months of age and 50% of children within six years of age have at least one episode of wheezing. Wheezing in young children can have a different etiology: it can be due to an underlying disease such as airway malformation, internal or external airway narrowing, and cystic fibrosis, or it can occur without an underlying disease.

In the latter case, the viral infection represents one of the main causes of wheezing especially in children under five/six years of age. However, not all viral infections cause wheezing.Numerous studies have confirmed a correlation between viral infections and asthma exacerbations in both adults and children. Furthermore, new evidence suggests that viral respiratory infections in the early years of life are related to the medium- and long-term development of asthma There is ample clinical evidence demonstrating a link between early viral infections (especially RV and RSV) and the onset of asthma exacerbations.

In addition to the viruses mentioned above, enteroviruses, bocaviruses, parainfluenza viruses, coronaviruses, metapneumoviruses, influenza viruses and adenoviruses also seem to be implicated.

RSV (respiratory syncytial virus) is the most common cause of bronchiolitis in the first year of life, causes hospitalization and typically circulates in temperate climates from November to April with peaks in the winter months

Although RSV has long been identified as the leading cause of childhood bronchiolitis, the use of molecular techniques, such as PCR, has also identified rhinovirus as a causative agent of asthma exacerbations. Rhinovirus, which circulates year-round with peaks during the fall and spring, as well as being a cause of upper respiratory tract infections, has been shown in some clinical investigations to infect the lower airways, to be associated with childhood bronchiolitis and become a dominant pathogen in wheezing disease as children get older.

In the search for new therapeutic and prevention alternatives that can be considered a valid contribution to reduce the effects of viral infection, the focus has been on effective and early treatments to help prevent the spread of the virus or to neutralize viruses at an early stage when they are lodged in the upper respiratory tract and therefore in the nose, since this is the probable and first route of entry for viruses and therefore for infections.

A nasal spray based on resveratol and carboxymethylbetaglucan (Linfovir® plus nasal spray) was therefore considered, which could be useful in hindering the entry of pathogens (viruses and bacteria) into the nasal cavities thanks to the mechanical action of the washing which goes to counter the engraftment and the consequent easier proliferation of the virus. Furthermore, the product contains resveratrol, a substance of natural origin, produced by various plants in response to stress or injury induced by microorganisms or environmental hazards which protects fruit and vegetables from fungal infections. This plant extract has been widely recognized as having antioxidant properties capable of counteracting the inflammatory stages associated with pathologies of the rhinosinusal tract. Patients infected with respiratory viruses, in fact, show an increased inflammatory state, with high levels of pro-inflammatory cytokines, such as tumor necrosis factor (TNF)α, interleukin IL-6, IL-8 and interferons, in the nasopharyngeal fluids and in plasma. Additionally, in severe viral infections, reactive oxygen species (ROS) produced by inflammatory cells, such as polymorphonuclear cells and neutrophils, recruited to the site of inflammation lead to lung damage.

On the basis of these assumptions, an interventional, randomized, multicenter and controlled clinical study was designed to evaluate whether the spray solution, used to hydrate and clean the nasal mucous membranes at a dosage of 2 sprays per nostril, 2 times a day (in prevention) and 2 sprays per nostril, 4 times a day (in the acute phase), is safe and effective in preventing and treating viral infections typical of the autumn/winter season in preschool wheezing children particularly prone to infections and asthma exacerbations. Thanks to the mechanical effect of washing and through the antioxidant and anti-inflammatory efficacy of resveratrol, amply demonstrated in vitro, the Investigators will evaluate, in the present study, whether the topical administration of resveratrol at the level of the nasal district, in the form of a nasal spray, is able to reduce the number of days in which preschool children present symptoms attributable to respiratory infections.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with wheezing

  * Patients aged between 3 and 6 years (inclusive) at the time of enrollment of both genders
  * Signature of the informed consent
  * Availability of a mobile phone capable of installing VIR@PP

Exclusion Criteria:

* Inability to adequately understand the Italian language
* Presence of autoimmune pathologies, immunodeficiency, neuromuscular diseases, congenital cardiomyopathies, metabolic diseases
* Presence of other syndromes and genetic pathologies
* Patients on therapy with other drugs (steroids for topical and/or oral use)
* Abnormalities of the nose or other conditions (e.g. severe hypotonia etc…) which make the administration of a nasal spray impossible or unsafe
* Denial of informed consent
* Participation in other clinical studies

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 252 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of the number of days with respiratory symptoms compared to placebo | 3 months
  To determine whether taking resveratrol in the form of a nasal spray changes the number of days with respiratory symptoms compared to placebo.

SECONDARY OUTCOMES:
In case of exacerbations, verify the change in the number of respiratory exacerbations and their duration of the group treated with resveratrol in the form of nasal spray vs the control group. | 3 months
  In case of exacerbations, verify the change in the number of respiratory exacerbations and their duration of the group treated with resveratrol in the form of nasal spray vs the control group. The number of days of use of antipyretics, oral corticosteroids and salbutamol will also be evaluated in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Miraglia del Giudice, Prof., Principal Investigator — University of Campania Luigi Vanvitelli - Naples; Italy 80138
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No